CLINICAL TRIAL: NCT05184777
Title: Evaluation of Salivary ELISA for Hormone Monitoring in IVF Patients
Acronym: SALIVA_MINT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Collaborators: MINT DIAGNOSTICS (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2107-VLC-071-EB
Record Dates: First submitted 2021-12-22; First posted 2022-01-11 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Infertility, Female; Reproductive Sterility
Keywords: ELISA; Saliva; Progesterone; Oestradiol; Early follicular phase; Mild follicular phase; Late follicular phase
MeSH Terms: conditions — Infertility, Female; Infertility

STUDY DESIGN:
Intervention Model Description: Prospective unicentric study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients undergoing ovarian stimulation for IVF/ICSI (Experimental): 90 patients undergoing ovarian stimulation for IVF/ICSI; Low, average and high responders will be included in equal proportions, in order to cover the widest range of hormonal values (30 blood and saliva samples per ovarian stimulation point will be taken for determination of progesterone and oestradiol).
  Interventions: Diagnostic Test: Determination of progesterone and oestradiol
- Patients for embryo transfer (ET) undergoing hormonal replacement therapy (Experimental): 30 patients for embryo transfer (ET) undergoing hormonal replacement therapy. These patients will only have a progesterone determination in their blood and saliva samples on the day of ET.
  Interventions: Diagnostic Test: Determination of progesterone and oestradiol

INTERVENTIONS:
Diagnostic Test: Determination of progesterone and oestradiol — Blood and saliva samples will be taken for determination of progesterone and oestradiol hormones.

SUMMARY:
In assisted reproductive treatment (ART), it is necessary to follow closely the stimulation cycles of patients undergoing these treatments in order to monitor the number and size of developing follicles. Oestradiol (E2) and progesterone (P) are products of steroidogenesis and the concentrations of both hormones increase with the diameter of the growing follicle and accurate and reliable methods to measure E2 and P are essential to assess treatment response and support clinical decision. Measurement of both hormones, as well as monitoring of follicle growth through ultrasound measurements, is an important part of ovarian stimulation, requiring patients to undergo multiple blood draws. It is often a physically and emotionally painful process and the most convenient solution to this problem is the measurement of hormone concentration in other biological fluids. Salivary diagnostic tests are a less invasive, inexpensive and stress-free alternative to measurements of hormone concentration in other biological fluids. The current study pretends to evaluate the correlation between salivary ELISA assays and serum determination of progesterone and oestradiol concentrations IVF patients. In addition, secondary objectives include the measurement of diurnal variability of salivary hormone levels and patient experience with saliva collection as users.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing IVF/ICSI treatment
* Patients planned to embryo transfer (ET) undergoing hormonal replacement therapy
* Aged from18-45 years old.
* BMI 19-30 kg/m2
* Signed written informed consent

Exclusion Criteria:

• Patients suffering for any systemic disease or endocrine disorder will be excluded foe the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2022-02-03 (Actual); Primary Completion 2022-05-17 (Actual); Study Completion 2023-02-20 (Actual)

PRIMARY OUTCOMES:
To evaluate the correlation between salivary ELISA assays and serum determination of progesterone and oestradiol concentrations IVF patients. | 12 months
  between salivary ELISA assays and serum determination of progesterone and oestradiol concentrations

SECONDARY OUTCOMES:
Diurnal variability of salivary progesterone and oestradiol levels | 12 months
  Measurement of progesterone and oestradiol levels
Patient User Experience with saliva collection | 12 months
  Registry of patient experience with saliva collection as users using a specific questionary. (Yes/No question)

CONTACTS AND LOCATIONS:
Locations (1):
- IVI Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No